CLINICAL TRIAL: NCT00215787
Title: Investigation of the Association Between Nasal Polyposis and Extraesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Head and Neck Surgery Associates (Other)
Responsible Party: Scott Phillips MD, Head and Neck Surgery Associates
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0165
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Results first posted 2010-09-22 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Nasal Polyps; Gastroesophageal Reflux
Keywords: Nasal polyps; Gastroesophageal Reflux
MeSH Terms: conditions — Nasal Polyps; Gastroesophageal Reflux | interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lansoprazole — Lansoprazole 30 mg BID for 1 year
  Other Names: Prevacid is the brand name for this drug

SUMMARY:
Although nasal polyposis has been recognized as an inflammatory process for many years, the true etiology of nasal polyposis mainly unknown. Despite surgical removal, the recurrence rate after surgery has been reported as high as 87% within the first year after surgery. Anecdotally the Principal Investigator found an incidence of pH probe-proven laryngopharyngeal reflux approaching 80% in his patients with nasal polyposis. Although his number of cases was small, the incidence of recurrence of polyps in these patients was 17%.

The PI believes that such an association is too great to be explained by chance alone, and deserves further study. He anticipates two contributions to the literature from this study, the first documenting the incidence of extraesophageal (laryngopharyngeal) reflux in patients with polyposis, and the second showing the impact of reflux treatment on the recurrence rate of the polyps, initially after one year of therapy.

DETAILED DESCRIPTION:
Although nasal polyposis has been recognized as an inflammatory process for many years, the true etiology of nasal polyposis mainly unknown. Despite surgical removal, the recurrence rate after surgery has been reported as high as 87% within the first year after surgery. Anecdotally the Principal Investigator found an incidence of pH probe-proven laryngopharyngeal reflux approaching 80% in his patients with nasal polyposis. Although his number of cases was small, the incidence of recurrence of polyps in these patients was 17%.

The PI believes that such an association is too great to be explained by chance alone, and deserves further study. He anticipates two contributions to the literature from this study, the first documenting the incidence of extraesophageal (laryngopharyngeal) reflux in patients with polyposis, and the second showing the impact of reflux treatment on the recurrence rate of the polyps, initially after one year of therapy.

Eligible patients found to have nasal polyps will be offered the chance to participate in this study. They will undergo non-invasive pH probe monitoring for 24 hours. If extraesophageal (laryngopharyngeal) reflux is discovered, they will be provided (at no cost) proton pump inhibitor medication (PPI), prescribed in accordance with published standards in the otolaryngology literature. Their polyposis will be treated as any other patient presenting with polyposis; participation in the study will not affect the course of polyp treatment. The incidence of recurrence will be monitored and recorded over the first year after treatment.

Included: Subjects will be adults with nasal polyposis, recruited from the PI's private practice, will not be currently taking a PP!, will be able and willing to undergo a noninvasive 24 hour pH probe study, and willing to take a PPI. Excluded: patients who are pregnant, have a history of surgical treatment for reflux disease, history of allergic or adverse reaction to Prevacid or adverse reaction to Prevacid during the study period, and those not meeting inclusion criteria.

In addition to routine office otolaryngology examination, subjects will undergo noninvasive 24 hour esophageal pH probe monitoring. The probe is swallowed and placed in the same manner as a feeding tube. The procedure is done in the office. No sedation is required, but the mucosa may be sprayed with topical 4% lidocaine for comfort. This procedure is the standard for diagnosis of extraesophageal (laryngopharyngeal) reflux, and will be performed in accordance with manufacturer guidelines

Risks include temporary dysphagia while the probe is in place, and nasal irritation. Mild, self-limited epistaxis has been rarely reported

The procedure will be done within manufcturer guidelines under direct vision. Topical Afrin may be used to control any mild epistaxis. Topical 4% lidocaine will be applied to minimize dysphagia. These steps have proven very affective in minimizing these risks.

If the study hypothesis is correct, the patient may have an diminished risk of recurrence of their nasal polyposis. If the patient is found to have previously undiagnosed reflux disease, this will allow it to be treated appropriately. Undiagnosed/untreated reflux has been associated with multiple medical problems including laryngeal and esophageal cancer. The patient will be given their PPI medication free of charge for the duration of the study. The noninvasive pH probe study will be done free of charge. No direct monetary payment will be given to participants.

ELIGIBILITY:
Inclusion Criteria:

Subjects will:

* Be adults with nasal polyposis
* recruited from the PI's private practice
* Not be currently taking a PPI
* Be able and willing to undergo a noninvasive 24 hour pH probe study; and
* Take a PPI.

Exclusion Criteria:

Patients who:

* Are pregnant
* Have a history of surgical treatment for reflux disease
* History of allergic or adverse reaction to Prevacid or adverse reaction to Prevacid during the study period; and
* Do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Phillips, MD, Principal Investigator — Head and Neck Surgery Associates
Locations (1):
- Head and Neck Surgery Associates, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Vento SI, Ertama LO, Hytonen ML, Wolff CH, Malmberg CH. Nasal polyposis: clinical course during 20 years. Ann Allergy Asthma Immunol. 2000 Sep;85(3):209-14. doi: 10.1016/S1081-1206(10)62468-4. PMID 11030275
- [Background] Virolainen E, Puhakka H. The effect of intranasal beclomethasone dipropionate on the recurrence of nasal polyps after ethmoidectomy. Rhinology. 1980 Mar;18(1):9-18. PMID 6988929
- [Background] Postma GN, Johnson LF, Koufman JA. Treatment of laryngopharyngeal reflux. Ear Nose Throat J. 2002 Sep;81(9 Suppl 2):24-6. PMID 12353429

RESULTS

PARTICIPANT FLOW:
Groups:
- Lansoprazole: Lansoprazole 30mg BID for one year
Period: Overall Study
Arm/Group | Lansoprazole
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lansoprazole
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Presence of Reflux in Patients With Polyposis
Description: Presence of Laryngopharyngeal reflux was measured by 24 hour pH impedance probe monitor per equipment manufacturer software. Two or more episodes in twenty four hours was considered positive, in accordance with published standards.
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 20
participants | 15

ADVERSE EVENTS:
Description: Serious and non-serious adverse events were not assessed.
Arm/Group | Lansoprazole
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes